CLINICAL TRIAL: NCT03564301
Title: Metronidazole as an Adjunct of Non- Surgical Treatment of Peri-implantitis : a 6-months Placebo- Controlled Clinical Trial in Humans
Brief Title: Metronidazole as an Adjunct of Non- Surgical Treatment of Peri-implantitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan Blanco Carrión (Other)
Collaborators: Osteology Foundation (Other)
Responsible Party: Sponsor-Investigator, Juan Blanco Carrión, Principal investigator, University of Santiago de Compostela
Organization: University of Santiago de Compostela (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APB-MET-2017-01
Record Dates: First submitted 2018-05-19; First posted 2018-06-20 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-03

CONDITIONS: Peri-Implantitis
Keywords: Peri-implantitis; antibiotics; Metronidazole; non- surgical treatment
MeSH Terms: conditions — Peri-Implantitis | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: PLACEBO-CONTROLLED CLINICAL TRIAL IN HUMAN
Who Masked: Participant, Care Provider, Investigator
Masking Description: It will not be possible to know which patient will correspond the prescription of the antibiotic or the placebo until the end of treatment. One of the researchers will be masked and will deliver the boxes with the placebo or the antibiotic according to the result of randomization. He will be different from the researcher who perform the treatment. This means that the treatment group will be masked to patients and dentists.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronidazole 250mg (Active Comparator): Systemic antibiotic: Metronidazole 250mg , 2 capsules three times a day, for 7 days.
  Interventions: Drug: Metronidazole 250 MG
- Placebo (Placebo Comparator): Placebo: same shape, size and dosis as test
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Placebo oral capsule — Immediately after the end of non surgical treatment of periimplantitis and depending on the result of randomization, the exact number of tablets of the placebo to be taken during the following days will be given to the patient.
  Arms: Placebo
Drug: Metronidazole 250 MG — Immediately after the end of non surgical treatment of periimplantitis and depending on the result of randomization, the exact number of tablets of the antibiotic to be taken during the following days will be given to the patient.
  Arms: Metronidazole 250mg

SUMMARY:
The use of systemic antibiotics as and adjunct to non-surgical peri-implant therapy may be an improvement in comparison to these therapies alone. The primary objective is the evaluation of significant changes in probing pocket depth between non-surgical with or without antibiotics.

This is a controlled-placebo clinical trial design. Patients with osseointegrated oral implants will be selected and recruited from a university clinic. Oral hygiene instruction and non-surgical debridement at implants will be provided with ultrasonic devices and immediately after, patients will be prescribed:

Group Control: A placebo with the same characteristics as the antibiotic Group Test: Systemic antibiotics (Metronidazole 250mg, 2 capsules three times a day, for 7 days Three and six months after non-surgical treatment, clinical parameters will be registered and radiographs compared using reproducible landmarks. Any adverse event will be also recorded.

DETAILED DESCRIPTION:
Microbial colonization of implant surface is the main causative factor of periimplantitis. Non-surgical treatment have been shown to be ineffective in bacterial control. The capacity of certain bacteria to invade soft tissues in periodontal lesions and a possible invasion in peri-implant diseases, could also be a good reason. Mombelli and Lang in a case-series study observed a significant reduction on probing depths and microbial parameters after non-surgical treatment and systemic antimicrobial therapy (ornidazole) of implants affected by marked loss of bone.

The rationale for conducting this research is to demonstrate that there may be significant differences in clinical, radiographic and microbiological parameters if systemic metronidazole is prescribed in conjunction with non-surgical treatment of peri-implantitis lesions. If there are differences, and a further improvement is observed in evaluated parameters, treatment protocols for these prevalent lesions could have been modified.

The objective of this research is to check whether there are differences in clinical, radiographic and microbiological parameters when performing non-surgical treatment to treat peri-implantitis with adjunctive administration of systemic metronidazole or a placebo.

Design: This research is designed as a parallel group, placebo-controlled, randomized, double-blind clinical study.

Population: Patients who come to the Periodontology Department, Faculty of Dentistry, University of Santiago de Compostela with dental implants presenting pathology.

Treatment Groups: Study group: patients treated by non-surgical treatment in conjunction with systemic metronidazole.Control group: patients treated by non-surgical treatment in conjunction with a placebo.

Randomization:After checking the inclusion criteria, signing the informed consent and included in the study. All subjects will be randomly assigned a number and one of the treatment group. The randomization will be done by a computer program for a simple randomization assignment.

Treatment: Non-surgical treatments will be performed under local anaesthesia . In cases where the prosthesis is screwed and screw access is possible, it will be removed during treatment and re-placed once completed. The patient will rinse with a mouthwash of chlorhexidine digluconate 0.12% and then implants affected will be debrided by ultrasound and manual curettes with the objective of removing deposits of plaque and calculus that are attached to the surface of the implant or prosthesis. Once the debridement is finished, pockets will be irrigated with chlorhexidine for 2 minutes and the surface of the prostheses polished using rubber cups and polishing paste.Immediately after the end of treatment and depending on the result of randomization, the exact number of tablets of the antibiotic or placebo to be taken during the following days will be given to the patient. The patient will be instructed in oral hygiene with either manual or electric toothbrush and interdental hygiene at the time of the completion of treatment. Subsequently, at 4 weeks, motivation and hygiene instructions will be strengthened by modifying brushing technique when deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Presence of at least 1 implant diagnosed with peri-implantitis (Presence of BOP and/or suppuration, with 2 mm of detectable bone loss after initial remodeling, and PD≥ 4 mm as defined by Daubert et al. 2015).
* Absence of implant mobility.
* History of taking systemic antibiotics in the preceding 3 months.
* No systemic pathology that contraindicated the completion of treatment.
* The patient understands the treatment and willing to comply.
* The patient is willing to give written informed consent and can do

Exclusion Criteria:

* Pregnant.
* Metronidazole allergies
* Patients on treatment with bisphosphonates.
* Uncontrolled periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-03 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Change in probing depth | baseline, 2 and 6 months after treatment
  Probing depth is the distance from the gingival margin to the bottom of the periodontal pocket (junctional epithelium). It is measured with a millimetric probe CP15 Hu-Friedy UNC at six points in each implant (mesial, distal and medial in buccal and lingual).

SECONDARY OUTCOMES:
Recession | baseline, 2 and 6 months after treatment
  the distance is measured from the free gingival margin (more coronal portion of the free gingiva) to the cement enamel junction. The following values are obtained:
  * Zero: if the level of the cement enamel junction.
  * Negative: the free gingival margin is apical to the cement enamel junction.
  * Positive: when the free gingival margin is coronal to the cement enamel junction.
Attachment level | baseline, 2 and 6 months after treatment
  Distance from the cement enamel junction to the bottom of the periodontal pocket (probing depth + recession).
Bleeding Index | baseline, 2 and 6 months after treatment
  it will be recorded in six locations per tooth. It will be registered as presence or absence. If bleed- ing occured within 10-15 s, a positive score will be given.
Peri-implant bone loss. | baseline, 2 and 6 months after treatment
  Distance from the implant shoulder to the first bone-implant contact in mesial and distal aspects of each implant.. The extent of peri-implant bone loss will be performed with Kodak® software and a correction of the vertical distortion of the x- rays will be done by the technique described by Tonetti et al. (1993).
Microbiological variable | baseline and 6 months after treatment
  in terms of presence of periodontal pathogens and bacterial load. Deeper locations around each implant will be selected. The samples will be analyzed by real-time PCR. It will be recorded as the total percentage of each bacterium
plaque index | baseline, 2 and 6 months after treatment
  it will be recorded in four locations per tooth. It will be registered as presence or absence. Plaque present along the gingival margin that could be easily removed with the tip of a probe was recorded. Percentage scores for the presence of plaque over all examined sites will be calculated for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of periodontology, faculty of Odontology, Santiago de Compostela, Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carcuac O, Derks J, Charalampakis G, Abrahamsson I, Wennstrom J, Berglundh T. Adjunctive Systemic and Local Antimicrobial Therapy in the Surgical Treatment of Peri-implantitis: A Randomized Controlled Clinical Trial. J Dent Res. 2016 Jan;95(1):50-7. doi: 10.1177/0022034515601961. Epub 2015 Aug 18. PMID 26285807
- [Result] Mombelli A, Lang NP. Antimicrobial treatment of peri-implant infections. Clin Oral Implants Res. 1992 Dec;3(4):162-8. doi: 10.1034/j.1600-0501.1992.030402.x. PMID 1298430
- [Result] Renvert S, Samuelsson E, Lindahl C, Persson GR. Mechanical non-surgical treatment of peri-implantitis: a double-blind randomized longitudinal clinical study. I: clinical results. J Clin Periodontol. 2009 Jul;36(7):604-9. doi: 10.1111/j.1600-051X.2009.01421.x. PMID 19538334
- [Result] Renvert S, Roos-Jansaker AM, Claffey N. Non-surgical treatment of peri-implant mucositis and peri-implantitis: a literature review. J Clin Periodontol. 2008 Sep;35(8 Suppl):305-15. doi: 10.1111/j.1600-051X.2008.01276.x. PMID 18724858
- [Result] Persson GR, Samuelsson E, Lindahl C, Renvert S. Mechanical non-surgical treatment of peri-implantitis: a single-blinded randomized longitudinal clinical study. II. Microbiological results. J Clin Periodontol. 2010 Jun;37(6):563-73. doi: 10.1111/j.1600-051X.2010.01561.x. PMID 20507380
- [Derived] Blanco C, Pico A, Dopico J, Gandara P, Blanco J, Linares A. Adjunctive benefits of systemic metronidazole on non-surgical treatment of peri-implantitis. A randomized placebo-controlled clinical trial. J Clin Periodontol. 2022 Jan;49(1):15-27. doi: 10.1111/jcpe.13564. Epub 2021 Oct 28. PMID 34713471
- See also: Mechanical non-surgical treatment of peri-implantitis: a single-blinded randomized longitudinal clinical study. II. Microbiological results — https://www.ncbi.nlm.nih.gov/pubmed/?term=Persson%2C+G.+Rutger%2C+Emelie+Samuelsson%2C+Christel+Lindahl%2C+and+Stefan+Renvert.+%22Mechanical+Non-surgica+Treatment+of+Peri-implantitis%3A+A+Single-blinded+Randomized+Longitudinal+Clinical+Study.+II.+Microbiological+Results.
- See also: Adjunctive Systemic and Local Antimicrobial Therapy in the Surgical Treatment of Peri-implantitis: A Randomized Controlled Clinical Trial. — https://www.ncbi.nlm.nih.gov/pubmed/26285807
- See also: Antimicrobial treatment of peri-implant infections — https://www.ncbi.nlm.nih.gov/pubmed/?term=Mombelli%2C+A.%2C+and+N.+P.+Lang.+%22Antimicrobial+Treatment+of+Peri-implant+Infections.%22
- See also: Mechanical non-surgical treatment of peri-implantitis: a double-blind randomized longitudinal clinical study. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Renvert%2C+Stefan%2C+Emelie+Samuelsson%2C+Christel+Lindahl%2C+and+Gösta.+Rutger+Persson.+%22Mechanical+Non-surgica+Treatment+of+Peri-implantitis%3A+A+Double-blind+Randomized+Longitudinal+Clinical+Study.+I%3A+Clinical+Results.
- See also: Non-surgical treatment of peri-implant mucositis and peri-implantitis: a literature review. — https://www.ncbi.nlm.nih.gov/pubmed/?term=Renvert%2C+Stefan%2C+Ann-Marie+Roos-Jansåker%2C+and+Noel+Claffey.+%22Non-surgical+Treatment+of+Peri-implant+Mucositis+and+Peri-implantitis%3A+A+Literature+Review.